CLINICAL TRIAL: NCT05549427
Title: A Retrospective Cohort Study on Ventilator Associated Pneumonia Caused by Multi-Drug Resistance Organism in SQUH ICU
Brief Title: Ventilator Associated Pneumonia by Multi-Drug Resistant Organism
Acronym: VAP-MDR
Status: Completed | Type: Observational
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Dr Jyoti Burad, Principle investigator, Sultan Qaboos University
Other Study IDs: MREC#2783
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Ventilator Associated Pneumonia; Multi-antibiotic Resistance
Keywords: Ventilator Associated Pneumonia; Multi drug resistance; antibiotics; length of stay; mortality
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ventilation — Ventilation in ICU

SUMMARY:
Ventilator-associated pneumonia (VAP) is an infection of the pulmonary parenchyma in patients exposed to invasive mechanical ventilation for at least 48 h and is part of ICU-acquired pneumonia. VAP is one of the most frequent ICU-acquired infections. Reported incidences vary widely from 5 to 40%, depending on the setting and diagnostic criteria. The estimated attributable mortality of VAP is around 10%. Investigators will focus this study on the current understanding of the epidemiology and treatment of VAP caused by multi-drug resistant (MDR) organisms. The MDR organisms are significant threats to the prognosis of the ICU patient. They are challenging to treat because of a limited number of newer antibiotics available for treatment. Understanding their distribution and sensitivity pattern may provide clues on how to deal with this significant problem. The current study examines the distribution of MDR organisms in VAP and its incidence and outcome. Investigators will also study the sensitivity pattern of these MDR organisms and how it affects the patient outcome. All patients admitted to adult ICU will be scanned, positive respiratory cultures will be noted, and those with VAP will be studied in detail. Patient data will be collected using the hospital information system.

DETAILED DESCRIPTION:
Introduction Ventilator-associated pneumonia (VAP) is defined as an infection of the pulmonary parenchyma in patients exposed to invasive mechanical ventilation for at least 48 h and is part of ICU-acquired pneumonia. VAP is one of the most frequent ICU-acquired infections. Reported incidences vary widely from 5 to 40%, depending on the setting and diagnostic criteria. VAP is associated with prolonged duration of mechanical ventilation and ICU stay. The estimated attributable mortality of VAP is around 10%.

Investigators will focus this study on the current understanding of the epidemiology and treatment of VAP caused by multi-drug resistant (MDR). Other conditions such as ventilator-associated tracheobronchitis are not detailed.

The MDR organisms are significant threats to the prognosis of the ICU patient. These organisms are usually acquired in hospitals due to multiple factors like antibiotic use, immunosuppression, prolonged stay in the hospital, etc. They are challenging to treat because of a limited number of newer antibiotics available for treatment. Understanding their distribution and sensitivity pattern may provide clues on how to deal with this significant problem.

Aim of the Study :

The current study examines the distribution of MDR organisms in VAP and its incidence and outcome.

The primary outcome is to find the distribution of MDR bacteria in VAP-positive patients

The secondary outcomes

1. is to find the incidence of VAP in ICU patients.
2. to find outcomes for VAP patients.
3. to study the antibiotic sensitivity for VAP-causing organisms.

Investigators hope to formulate improvement strategies to minimize the incidence of MDR VAP, enhance ICU care, and reduce the incidence of VAP in ICU.

Methodology

Study Population: General Adult (>13 years) ICU patients on ventilators at SQUH

Study Design and Methods:

Design: This is a single center retrospective cohort study.

Sample size: All ICU patients on ventilators fulfilling inclusion criteria during the study period starting from 1/04/2021 to 31/03/2022

Study Method:

After obtaining ethical approval, all the patients admitted to ICU during the study period will be scanned for eligibility criteria. Patients with VAP will be studied using electronic patient records (EPR).

Demographic Data: Age and gender of the patients will be recorded. Diagnosis Data: Positive respiratory culture for MDR, Treatment Data: Empirical antibiotics and treatment of VAP Microbiology data: sensitivity and culture reports Other data: VAP days, ventilator days, and outcome: extubation, tracheostomy, survival, death.

Justification of the current study:

In this study, Investigators intend to determine the incidence of VAP due to MDR organism and associated outcomes. This will help in understanding VAP due to MDR organisms.

Data Management and Analyses:

Statistical analysis: Database for the study sample shall be created in SPSS-23. Categorized variables shall be displayed as percentages using frequency tables and pie charts or bar charts, and continuous variables shall be shown as Mean ± SD and error bar charts.

To test the significance of association between categorized variables, Chi-square or Fisher's exact test, as appropriate, shall be used. To test the significance of the difference between the means of two groups, an independent sample t-test will be applied if the distribution pattern of the variable under study is normal, and in case of non-normal behavior of the data; the Mann-Whitney test shall be applied. Similarly, for comparing means of 3 or more groups, ANOVA or Kruskal-Wallis test shall be used depending on the distribution pattern of the study variable. A P-value of .05 or less shall be taken as significant.

The analysis results will be used in a suitable form for publication.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (more than 13 years old) admitted to ICU (covid/non-covid) (for VAP rate)
* Patient who got intubation and mechanical ventilation for more than 48 hours (for VAP0
* Positive MDR bacterial respiratory culture for defining MDR VAP

Exclusion Criteria for MDR VAP:

* Non-ventilated patients.
* Patient with tracheobronchitis
* Patients positive for fungal cultures
* Patients with pneumonia before intubation
* Non-MDR VAP

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients (>13 years) admitted to ICU on a ventilator at a tertiary level center were scanned. Those who developed VAP with MDR organism (after 48 hours of ventilation and with new cultures after the initial negative culture) were labeled as MDR VAP cases. The remaining ventilated patients were considered to calculate VAP rate.
Sampling Method: Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Distribution of Multi-Drug Resistant (MDR) bacteria in VAP positive patients | upto 90 days
  Frequency and classes of MDR organisms isolated from respiratory specimens of ventilated patients for more than 48 hours

SECONDARY OUTCOMES:
Incidence of MDR-VAP in ICU patients | upto 90 days
  Incidence of VAP with MDR organisms during the study period.
Outcome of MDR-VAP patients | upto 90 days
  Outcomes like: Survival versus Mortality and Extubation versus Tracheostomy
Antibiotic sensitivity for MDR-VAP causing organism | upto 90 days
  The antibiotic sensitivity of MDR-VAP organisms

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Burad, MD, EDIC, Principal Investigator — Sultan Qaboos University Hospital
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared with those who ask for it by email to the principal investigator for the research. The patient data and the statistical plan will be shared
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after three months of publication of the present study indefinitely.
Access Criteria: Those who require data for research, will be provided with this dataset.
URL: https://data.mendeley.com/

REFERENCES:
- [Background] Djordjevic ZM, Folic MM, Jankovic SM. Distribution and antibiotic susceptibility of pathogens isolated from adults with hospital-acquired and ventilator-associated pneumonia in intensive care unit. J Infect Public Health. 2017 Nov-Dec;10(6):740-744. doi: 10.1016/j.jiph.2016.11.016. Epub 2017 Feb 8. PMID 28189513
- [Background] Patil HV, Patil VC. Incidence, bacteriology, and clinical outcome of ventilator-associated pneumonia at tertiary care hospital. J Nat Sci Biol Med. 2017 Jan-Jun;8(1):46-55. doi: 10.4103/0976-9668.198360. PMID 28250674
- [Background] Gupta R, Malik A, Rizvi M, Ahmed M, Singh A. Epidemiology of multidrug-resistant Gram-negative pathogens isolated from ventilator-associated pneumonia in ICU patients. J Glob Antimicrob Resist. 2017 Jun;9:47-50. doi: 10.1016/j.jgar.2016.12.016. Epub 2017 Apr 10. PMID 28288860
- [Background] Grasselli G, Scaravilli V, Mangioni D, Scudeller L, Alagna L, Bartoletti M, Bellani G, Biagioni E, Bonfanti P, Bottino N, Coloretti I, Cutuli SL, De Pascale G, Ferlicca D, Fior G, Forastieri A, Franzetti M, Greco M, Guzzardella A, Linguadoca S, Meschiari M, Messina A, Monti G, Morelli P, Muscatello A, Redaelli S, Stefanini F, Tonetti T, Antonelli M, Cecconi M, Foti G, Fumagalli R, Girardis M, Ranieri M, Viale P, Raviglione M, Pesenti A, Gori A, Bandera A. Hospital-Acquired Infections in Critically Ill Patients With COVID-19. Chest. 2021 Aug;160(2):454-465. doi: 10.1016/j.chest.2021.04.002. Epub 2021 Apr 20. PMID 33857475
- [Background] Sangale A, Vivek B, Kelkar R, Biswas S. Microbiology of Ventilator-associated Pneumonia in a Tertiary Care Cancer Hospital. Indian J Crit Care Med. 2021 Apr;25(4):421-428. doi: 10.5005/jp-journals-10071-23790. PMID 34045810
- [Background] Papazian L, Klompas M, Luyt CE. Ventilator-associated pneumonia in adults: a narrative review. Intensive Care Med. 2020 May;46(5):888-906. doi: 10.1007/s00134-020-05980-0. Epub 2020 Mar 10. PMID 32157357